CLINICAL TRIAL: NCT04025502
Title: A Multi-Center Study of Event-Related Potential (ERP) Biomarkers in Subjects With Schizophrenia and Healthy Volunteer Subjects
Brief Title: Event-Related Potential (ERP) Biomarkers in Subjects With Schizophrenia and Healthy Volunteer Subjects
Status: Completed | Type: Observational
Sponsor: ERP Biomarker Qualification Consortium (Industry)
Collaborators: Novartis (Industry); Alkermes, Inc. (Industry); Anavex Life Sciences Corp. (Industry); Merck Sharp & Dohme LLC (Industry); Takeda (Industry); Sage Therapeutics (Industry); H. Lundbeck A/S (Industry); Astellas Pharma Inc (Industry); Apex Innovative Sciences (Unknown); Columbia University (Other); COGNISION (Unknown)
Responsible Party: Sponsor
Other Study IDs: EBS-A
Record Dates: First submitted 2019-06-23; First posted 2019-07-19 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
Keywords: ERP; EEG; Event-related potential; MMN; Schizophrenia; Electroencephalogram; Mismatch Negativity; N100; P3a; P3b
MeSH Terms: conditions — Schizophrenia | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva drug screen to rule out illicit drug use for all three visits (Screening visit, Baseline visit, and Retest visit).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer Subjects (HV): Male and female subjects 21-50 years of age, who are in good and stable health with no history or evidence of clinically relevant medical or neuropsychiatric illness.
  Healthy Volunteer Subjects will undergo Event-Related Potential (ERP)/electroencephalogram (EEG) testing with the COGNISION® System.
  Interventions: Device: Event-Related Potentials (ERP) and Electroencephalogram (EEG) testing with the COGNISION® System
- Subjects with Schizophrenia (SZ): Otherwise healthy male and female subjects 21-50 years of age, who have a current diagnosis of Schizophrenia with a duration of illness greater than or equal to one year.
  Subjects with Schizophrenia (SZ) will undergo Event-Related Potential (ERP)/electroencephalogram (EEG) testing with the COGNISION® System.
  Interventions: Device: Event-Related Potentials (ERP) and Electroencephalogram (EEG) testing with the COGNISION® System

INTERVENTIONS:
Device: Event-Related Potentials (ERP) and Electroencephalogram (EEG) testing with the COGNISION® System — The testing protocol consists of an auditory oddball Event-Related Potential (ERP) paradigm, 40Hz ASSR, and the collection of 6 minutes of resting electroencephalogram (EEG). During the ERP paradigm a variety of auditory stimuli are played through the system's earphones while voltage potentials are recorded from the subject's scalp. At the end of the ERP session, 6 minutes of EEG data will be recorded while the subject is resting. The entire procedure, including set up, instructions to the subject and actual test is expected to take 60-75 minutes.

SUMMARY:
This is an observational, non-interventional study that will recruit Healthy Volunteers (HV) and subjects with clinically confirmed Schizophrenia (SZ). The purpose of this study is to establish the mean and variance across the HV and SZ cohorts, sites, and repeated tests of the electroencephalogram(EEG)/Event-related potentials (ERP) measures.

DETAILED DESCRIPTION:
Among the most replicated pathophysiological findings in schizophrenia is the impairment of Event-Related Potentials (ERPs) recorded during the auditory oddball procedure. In this procedure, time-locked electroencephalogram (EEG) responses are recorded during auditory processing of frequent and rare tones differing in pitch or duration. In addition, a smaller but substantial literature has reported deficits in the auditory steady-state EEG response (ASSR) to a 40 Hz train of auditory tones in subjects with schizophrenia versus healthy control subjects.

While measurement of ERPs in the drug development setting has shown promise, the instruments, infrastructure, and standardization of these methods has lagged. New, portable, easy-to-use, Food and Drug Administration (FDA)-approved devices are now available for the automated collection and analysis of EEG and ERP data.

This observational, non-interventional, clinical study will recruit healthy volunteer subjects (HV) and subjects with clinically confirmed schizophrenia (SZ), and will establish the mean and variance across HV and SZ cohorts, sites and repeated tests, of EEG and ERP measures collected with a standardized EEG/ERP device. The study will also examine the relationship between specific EEG/ERP features and measures of positive, negative, and cognitive symptoms and global function in SZ subjects.

The data collected in this study is intended to replicate published observations of the magnitude of deficit in ERPs in SZ versus HV subjects, and to support the design of subsequent interventional studies that will make use of ERPs. Furthermore, these data will be submitted to support qualification of the ERP biomarkers through the FDA Drug Development Tools Biomarker Qualification Program.

ELIGIBILITY:
* Inclusion Criteria for Healthy Volunteer Subjects (HV)

  * Healthy male and female subjects 21-50 years of age (inclusive).
  * Are not currently or have not participated in any other clinical studies within 30 days of Screening.
  * Ability to understand the requirements of the study, provide written informed consent, abide by the study procedures, and agree to return for the required assessments.
  * Subject is in good and stable health with no history or evidence of clinically relevant medical or neuropsychiatric illness.
  * Fluent in English, even if English is not the primary language. Subjects must hold a U.S. citizenship only for eligibility to participate.
* Exclusion Criteria for Healthy Volunteer Subjects (HV)

  * Illicit drug use as determined by the saliva drug screen.
  * Current alcohol abuse as determined by the Investigator; or subject regularly consumed ≥3 alcoholic drinks/day during the 3 months prior to screening. One alcohol drink is approximately equivalent to: beer: 284 mL; wine: 125 mL (4 oz); or distilled spirits: 25 mL (1 oz).
  * Known (identifiable) biological family history of Schizophrenia spectrum disorders in a first or second degree relative.
  * Use of any first generation, sedating H1 antihistamines within 1 week prior to Screening or during the study. (see Medication Approval List)
  * Use of any sedative-hypnotic medications within 1 week prior to Screening or during the study. (see Medication Approval List)
  * Use of any other psychoactive medication known to interfere with ERP assessments within 1 week prior to Screening or during the study (see Medication Approval List).
  * Evidence or history of significant cognitive disorders, or other injuries, conditions, impairments, or situations that in the judgement of the Investigator would prevent safe and satisfactory completion of the study protocol.
  * Evidence or history of psychiatric illness as determined by the Mini International Neuropsychiatric Interview (MINI) for Psychotic Disorders.
  * Evidence of cognitive impairment as determined by performing ≥ 1.5 standard deviations lower compared to the age, sex, and education corrected mean on either the BACS Symbol Coding and/or Verbal Memory.
  * Significant intellectual disability as evidenced by a standardized WRAT-4 Reading Test standardized score < 70.
  * Unable to detect a 1000 and 2000 Hz tone at 40 dB in both ears.
  * Unable to tolerate the electrode cap for the duration of the testing session.
  * Known allergy to latex.
  * Use of products containing nicotine and/or caffeine 60 minutes prior to EEG/ERP testing.
* Inclusion Criteria for Subjects with Schizophrenia (SZ)

  * Otherwise healthy male and female subjects 21-50 years of age (inclusive).
  * Are not currently or have not participated in any other clinical studies within 30 days of Screening.
  * Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
  * Current diagnosis of schizophrenia.
  * Duration of schizophrenia illness ≥ 1 years.
  * Clinically stable and in the residual (non-acute) phase of their illness for at least 6 weeks prior to the study as evidenced by a stable medication regimen and no recent hospitalizations for acute Schizophrenia. The subject's clinical stability is ultimately up to the Investigator.
  * Maintained on a stable regimen of antipsychotic and/or permitted concomitant medications for at least 6 weeks prior to screening and during the study.
  * Subjects receiving treatment with up to 2, first or second-generation antipsychotics or other concomitant medications commonly prescribed to this patient population, may be included. (see Allowed Medications List)
  * Fluent in English, even if English is not the primary language. Subjects must hold a U.S. citizenship only for eligibility to participate.
* Exclusion Criteria for Subjects with Schizophrenia (SZ)

  * Illicit drug use as evidenced by the saliva drug screen.
  * Current alcohol abuse as determined by the Investigator; or subject regularly consumed ≥3 alcoholic drinks/day during the 3 months prior to screening. One alcohol drink is approximately equivalent to: beer: 284 mL; wine: 125 mL (4 oz); or distilled spirits: 25 mL (1 oz).
  * Use of any first-generation, sedating H1 antihistamines within 1 week prior to Screening or during the study (see Medication Approval List).
  * Use of any sedative-hypnotic medications within 1 week prior to Screening or during the study. (see Medication Approval List)
  * Use of any other psychoactive medication known to interfere with ERP assessments within 1 week prior to Screening or during the study (see Allowed Medications List).
  * Evidence or history of significant cognitive disorders, or other injuries, conditions, impairments, or situations that in the judgement of the Investigator would prevent safe and satisfactory completion of the study protocol.
  * Failure to confirm a diagnosis of Schizophrenia by the Investigator.
  * Significant intellectual disability as evidenced by a standardized WRAT-4 Reading Test score < 70.
  * Have no more than a moderate severity rating on hallucinations and delusions as evidenced by a PANSS items P1 ≥ 4 and P3 ≥ 4.
  * Have no more than a moderate severity rating on positive formal thought disorder as evidenced by a PANSS items G9 ≥ 4 and P2 ≥ 4.
  * Presence of more than minimal extrapyramidal symptoms as evidenced by a SAS score > 6.
  * Presence of more than minimal level of depressive symptoms as evidenced by a CDSS score ≥ 10.
  * Unable to detect a 1000 and 2000 Hz tone at 40 dB in both ears.
  * Unable to tolerate the electrode cap for the duration of the testing session.
  * Known allergy to latex.
  * Use of products containing nicotine and/or caffeine 60 minutes prior to EEG/ERP testing.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There will be four different sites where the participants will be selected in the following states: California, New Jersey, and New York.
  Recruitment methods:
  * Database of individuals who have agreed to be contacted
  * Advertisements
  * Physician to physician referrals
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Amplitude (in microvolts) for parameters from the ERP tests. | 12-18 months
  Amplitude (in microvolts) for the following parameters from the ERP tests will be collected as primary endpoints:
  1. Passive, Tone-deviant, Auditory Oddball ERP
     * N100
     * MMN
     * P3a
  2. Passive, Duration-deviant, Auditory Oddball ERP
     * N100
     * MMN
     * P3a
  3. Active, Auditory Oddball ERP
     * N100
     * P3b
Latency (in milliseconds) for parameters from the ERP tests. | 12-18 months
  Latency (in milliseconds) for the following parameters from the ERP tests will be collected as primary endpoints:
  1. Passive, Tone-deviant, Auditory Oddball ERP
     * N100
     * MMN
     * P3a
  2. Passive, Duration-deviant, Auditory Oddball ERP
     * N100
     * MMN
     * P3a
  3. Active, Auditory Oddball ERP
     * N100
     * P3b
Task accuracy from the behavioral response during the active, auditory oddball ERP test. | 12-18 months
  Task accuracy as a percentage of correct behavioral responses during the active, auditory oddball ERP test will be collected as a primary endpoint.
Reaction time from the behavioral response during the active, auditory oddball ERP test. | 12-18 months
  Reaction time for the correct behavioral responses to the test measured in milliseconds will be collected as a primary endpoint during the active, auditory oddball ERP test.
Total Power from the auditory steady-state response (ASSR) paradigm. | 12-18 months
  Total Power (measured in µv2/Hz) will be collected during the ASSR paradigm as a primary endpoint.
Inter-trial coherence (ITC) from the auditory steady-state response (ASSR) paradigm. | 12-18 months
  Inter-trial coherence (ITC) measured on a scale between 0 (no coherence) and 1 (maximum coherence) will be collected during the ASSR paradigm as a primary endpoint.
Absolute Power for Pharmaco-EEG parameters per IPEG guidelines. | 12-18 months
  Absolute Power (measured in µv2/Hz) will be collected from the Resting State EEG as a primary endpoint for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
  * Gamma power
Relative Power for Pharmaco-EEG parameters per IPEG guidelines. | 12-18 months
  Relative Power measured on a scale from 0 (no power in frequency band) to 1 (all EEG power in that frequency band) will be collected from the Resting State EEG as a primary endpoint for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
Dominant frequency in the Alpha frequency band per IPEG guidelines | 12-18 months
  Dominant frequency measured in Hz in the frequency interval between 6.0 and < 12.5 Hz will be collected from the Resting State EEG as a primary endpoint.
Theta/Beta ratio and Slow Wave index per IPEG guidelines. | 12-18 months
  Theta/Beta ratio and Slow Wave index (Alpha/Delta+Theta) measured in percentage will be collected from the Resting State EEG as primary endpoints.
Functional assessments as derived from the Brief Assessment of Cognition in Schizophrenia (BACS). | 12-18 months
  The following parameters will be collected for the BACS:
  BACS Variable Ranges Description Range Low Range High Unit Verbal Memory Total Score 0 75 n/a Digit Sequencing 0 28 n/a Token Motor Total Correct 0 100 n/a Verbal Fluency Total 0 100 n/a Symbol Coding 0 110 n/a Tower of London 0 22 n/a Verbal Memory T-Score -100 100 n/a Digit Sequencing T-Score -100 100 n/a Token Motor T-Score -100 100 n/a Verbal Fluency T-Score -100 100 n/a Symbol Coding T-Score -100 100 n/a Tower of London T-Score -100 100 n/a
Functional assessments as derived from the Positive and Negative Symptom Scale for Schizophrenia (PANSS). | 12-18 months
  The PANSS items are divided into three sections: Positive symptoms, negative symptoms, and general symptoms. The following parameters will be collected:
  PANSS Variable Ranges Description Range Low Range High Unit PANSS Items 1-30 1 7 n/a PANSS Total Score 30 210 n/a
Functional assessments as derived from the Virtual Reality Functional Capacity Assessment Tool (VRFCAT). | 12-18 months
  The following parameters for the VRFCAT will be collected:
  VRFCAT Variable Ranges Description Range Low Range High Unit VRFCAT- Adjusted Total Time 0 60000 msec VRFCAT- Total Error Count 0 60 n/a VRFCAT- Total Forced Progressions 0 12 n/a Adjusted Total Time T-Score -100 100 n/a Total Errors T-Score -100 100 n/a Total Forced Progressions T-Score -100 100 n/a

SECONDARY OUTCOMES:
Correlations between EEG/ERP measures and psychometric measures in Schizophrenia subjects. | 12-18 months
  Pearson Correlation coefficients between EEG/ERP measures and scores from the functional assessments (BACS, PANSS, and VRFCAT) will be collected as secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cecchi, PhD, Principal Investigator — ERP Biomarker Qualification Consortium
Locations (4):
- United States (4):
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Hassman Research Institute, Marlton, New Jersey
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jobert M, Wilson FJ, Ruigt GS, Brunovsky M, Prichep LS, Drinkenburg WH; IPEG Pharmaco-EEG Guidelines Committee. Guidelines for the recording and evaluation of pharmaco-EEG data in man: the International Pharmaco-EEG Society (IPEG). Neuropsychobiology. 2012;66(4):201-20. doi: 10.1159/000343478. Epub 2012 Oct 12. PMID 23075830
- [Background] Umbricht D, Krljes S. Mismatch negativity in schizophrenia: a meta-analysis. Schizophr Res. 2005 Jul 1;76(1):1-23. doi: 10.1016/j.schres.2004.12.002. Epub 2005 Jan 23. PMID 15927795
- [Background] Light GA, Hsu JL, Hsieh MH, Meyer-Gomes K, Sprock J, Swerdlow NR, Braff DL. Gamma band oscillations reveal neural network cortical coherence dysfunction in schizophrenia patients. Biol Psychiatry. 2006 Dec 1;60(11):1231-40. doi: 10.1016/j.biopsych.2006.03.055. Epub 2006 Aug 7. PMID 16893524
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Buchanan RW, Davis M, Goff D, Green MF, Keefe RS, Leon AC, Nuechterlein KH, Laughren T, Levin R, Stover E, Fenton W, Marder SR. A summary of the FDA-NIMH-MATRICS workshop on clinical trial design for neurocognitive drugs for schizophrenia. Schizophr Bull. 2005 Jan;31(1):5-19. doi: 10.1093/schbul/sbi020. Epub 2005 Feb 16. PMID 15888422
- [Background] Buchanan RW, Keefe RS, Umbricht D, Green MF, Laughren T, Marder SR. The FDA-NIMH-MATRICS guidelines for clinical trial design of cognitive-enhancing drugs: what do we know 5 years later? Schizophr Bull. 2011 Nov;37(6):1209-17. doi: 10.1093/schbul/sbq038. Epub 2010 Apr 21. PMID 20410237